CLINICAL TRIAL: NCT03356457
Title: Development of Agents to Diminish the Risk of Hypoglycemia-induced Brain Injury in Type 1 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2000029203
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hyperglycaemia (Diabetic)
MeSH Terms: conditions — Hyperglycemia | interventions — Dichloroacetic Acid

STUDY DESIGN:
Intervention Model Description: This will be a single center, placebo-controlled, cross-over, randomized clinical pilot study.
  At the screening visit informed consent will be obtained. Medical history and documents will be reviewed to screen potential subjects by inclusion and exclusion criteria. Subjects will receive a physical examination and laboratory blood work (BUN/creatinine, electrolytes, lipid profile, liver function, and HbA1c) as well as urine toxicology screens (to confirm self-report of alcohol, and drug information) to ensure good physical health.
Who Masked: Participant
Masking Description: Once stable hypoglycemia is reached, a cognitive testing battery will be administered by a study co-investigator who will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DCA in T1DM with severe hypoglycemia (Active Comparator): 12 T1DM subjects (C-peptide negative, HbA1c <7.5%) with a history of severe hypoglycemia and hypoglycemia unawareness as assessed by the Guy's and Thomas' Minimally Modified Clarke Hypoglycemia Survey, the Gold Score and the Edinburgh Hypoglycemia Survey and as evidenced by interview and glucose log and/or continuous glucose monitoring will receive a single dose of 12.5mg/kg dichloroacetate (DCA).
  Interventions: Drug: Dichloroacetate
- Placebo in T1DM with severe hypoglycemia (Placebo Comparator): 12 T1DM subjects (C-peptide negative, HbA1c <7.5%) with a history of severe hypoglycemia and hypoglycemia unawareness as assessed by the Guy's and Thomas' Minimally Modified Clarke Hypoglycemia Survey, the Gold Score and the Edinburgh Hypoglycemia Survey and as evidenced by interview and glucose log and/or continuous glucose monitoring will receive a placebo oral capsule.
  Interventions: Drug: Placebo oral capsule
- DCA in healthy control subjects (Active Comparator): 12 non-diabetic healthy subjects (fasting plasma glucose < 100 mg/dL, HbA1c < 6.0%), who are matched for age, gender, and weight to T1DM subjects, to serve as controls for the study. Each subject will receive a single dose of 12.5mg/kg dichloroacetate (DCA).
  Interventions: Drug: Dichloroacetate
- Placebo in healthy control subjects (Placebo Comparator): 12 non-diabetic healthy subjects (fasting plasma glucose < 100 mg/dL, HbA1c < 6.0%), who are matched for age, gender, and weight to T1DM subjects, to serve as controls for the study will receive a placebo oral capsule.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Dichloroacetate — Dichloroacetate is an isoform-unspecific inhibitor of four regulatory pyruvate dehydrogenase kinases, which are able to reduce entry of substrates into mitochondria by reducing the conversion of pyruvate to acetyl-CoA. Drug will be administered to subjects with sever hypoglycemia as well as healthy non-diabetic subjects.
  Other Names: DCA
  Arms: DCA in T1DM with severe hypoglycemia; DCA in healthy control subjects
Drug: Placebo oral capsule — A Placebo oral capsule identical in shape and color to those with active ingredient.
  Other Names: Placebo
  Arms: Placebo in T1DM with severe hypoglycemia; Placebo in healthy control subjects

SUMMARY:
To determine the effect of re-activation of brain glucose metabolism induced by dichloroacetate (DCA) on cognitive function and counterregulatory hormone responses in patients with type 1 diabetes (T1DM) with recurrent hypoglycemia.

DETAILED DESCRIPTION:
This will be a single center, placebo-controlled, cross-over, randomized clinical pilot study. The screening will take place at the Yale New Haven Hospital Research Unit (HRU) 10th floor, East Pavilion at 20 York St., New Haven, CT. At the screening visit informed consent will be obtained. Medical history and documents will be reviewed to screen potential subjects by inclusion and exclusion criteria. Subjects will receive a physical examination and laboratory blood work (BUN/creatinine, electrolytes, lipid profile, liver function, and HbA1c) as well as urine toxicology screens (to confirm self-report of alcohol, and drug information) to ensure good physical health.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Diagnosed C-peptide-negative T1DM, > 5 years duration, HbA1c of < 7.5%
* Intensive management, defined by frequent self-monitoring of glucose values and by the administration of 3 or more insulin injections each day (or the use of insulin pump therapy).
* History of severe hypoglycemia and hypoglycemia unawareness as assessed by the Guy's and Thomas' Minimally Modified Clarke Hypoglycemia Survey, the Gold Score and the Edinburgh Hypoglycemia Survey (see Appendix 1)
* Willingness to fast and to reduce insulin therapy for a limited time period

Group 2:

* Age, weight, and gender matched to group 1 subjects
* HbA1c <6%
* Good general health as evidenced by medical history and blood screening
* Willing to fast for a limited time period

Exclusion Criteria:

General criteria:

* Known allergic reactions to components of the study product(s)
* Participants carrying polymorphisms known to slow DCA metabolism (e.g. KGM or EGM allele [10])
* Treatment with another investigational drug or other intervention
* Active infection including hepatitis C, hepatitis B, HIV
* Any past or current history of alcohol or substance abuse
* Psychiatric or neurological disorders, including need for medications, including anxiolytics, and antidepressants
* Baseline Hgb < 10.5 g/dL in females, or < 12.5 g/dL in males. Blood donation within 30 days of the study
* History of coagulopathy or medical condition requiring long-term anticoagulant therapy (low-dose aspirin treatment is allowed)
* Co-existing cardiac, liver, and kidney disease
* Abnormal liver function tests
* GI disorders potentially interfering with the ability to absorb oral medications
* Women that are post-menopausal, pregnant (as assessed by pregnancy test that will be performed on female participants at reproductive age), or lactating.
* Any medical condition that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes
* Any medication assumed less than 30 days before the study sessions that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes.The list of medications to be avoided includes - but is not limited to - drugs known to influence metabolic and endocrine function (other than insulin in Group 1) and neuroactive medications.

Group 1:

* Detectable C-peptide;
* Untreated proliferative retinopathy;
* Creatinine ≥1.5 mg/dl, urinary albumin levels . 300 mg/day
* Autonomic neuropathy; painful peripheral neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
• Measurement of hormone changes during hypoglycemia | 1 day
  Plasma counterregulatory hormone concentrations will be collected during the controlled insulin-induced hypoglycemic portion of the study.

SECONDARY OUTCOMES:
cognitive function | 1 day
  Performance on a battery of cognitive tests assessing short term memory during controlled hypoglycemia. The Cantab battery of short-term memory tests will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States